CLINICAL TRIAL: NCT04832503
Title: Childhood Apraxia of Speech: Neurobiological and Behavioural Markers and Experience Dependent Changes of Neural Connectivity Induced by Treatment
Brief Title: Childhood Apraxia of Speech: Experience Dependent Changes Induced by Treatment
Acronym: CAS
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Anna Chilosi, MD, PhD Head of Neurolinguistic and Neuropsychological Research Laboratory. Coordinator of the Clinical Neuropsichological Unit, IRCCS Fondazione Stella Maris
Other Study IDs: RF-2016-02361560
Record Dates: First submitted 2021-02-20; First posted 2021-04-05 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Childhood Apraxia of Speech
Keywords: Treatment induced speech changes; PROMPT; MRI; Neuroplasticity
MeSH Terms: conditions — Apraxias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The PROMPT-treated group will include 12 children with idiopathic CAS. The pre-treatment assessment is aimed at evaluating the baseline speech and language level and at treatment planning. During a PROMPT session tactile-kinesthetic-proprioceptive inputs are consistently provided in order to shape speech movements, to give information on sequencing and timing, and to introduce constraints for the reduction of the degrees of freedom at the articulators' level in favour of motor control. In a PROMPT session the syllables, words and phrases are produced within a communicative context in play. Speech motor goals are, as soon as possible, integrated in goals for language and functional communication.
  Interventions: Behavioral: PROMPT- treatment
- GROUP 2: The LNSOM-treated group will include 12 children with idiopathic CAS. The pre-treatment assessment is aimed at evaluating the baseline speech and language level and at the treatment planning. None of the SLTs treating this group are PROMPT trained. According to the standard care methods used in Italy, the intervention consists of a linguistic and articulatory approach that includes auditory discrimination of phonemic categories at the syllable and word level and non-speech oral motor exercises. Receptive and expressive lexicon and morphosyntax are targeted depending on the children's linguistic profile.Differently from the PROMPT, selection of speech sounds to be targeted, is based on developmental speech sounds acquisition rather than motor criteria. According to this treatment approach, the motor goal is usually identified with the placement of the main articulator involved in the production of a speech sound.
  Interventions: Behavioral: LNSOM-treatment

INTERVENTIONS:
Behavioral: PROMPT- treatment — PROMPTs for Restructuring Oral Muscolar Phonetic Targets
  Groups: Group 1
Behavioral: LNSOM-treatment — Language Non-Speech Oral Motor Treatment
  Groups: GROUP 2

SUMMARY:
Childhood Apraxia of Speech (CAS) is a severe speech-language disorder whose aetiological, neuroanatomical correlates are largely unknown. Furthermore, little is known about the neuroplastic effects induced by different treatment approaches and their relationships with the potential changes in the speech behavioural features that express the core deficit of CAS.

Twenty four children with idiopathic CAS will be enrolled in a multidisciplinary study aimed at analysing the behavioural and neuroanatomical effects of a specific rehabilitative approach, PROMPT (PROMPTs for Restructuring Oral Muscular Phonetic Targets), that employs tactile-kinesthetic-proprioceptive cues vs a traditional speech-language treatment. The children will be allocated in two arms, one receiving a seven month cycle of individual PROMPT treatment, the other a traditional speech and language treatment for the same amount of time.The pre- and post-treatment speech and language performances and DTI and volumetric MR data will be compared in the two groups.

DETAILED DESCRIPTION:
Background: Childhood Apraxia of Speech (CAS) is a severe speech-language disorder whose etiological, neuroanatomical and genetic correlates are largely unknown. In this trial the effects of an innovative rehabilitative approach, PROMPT (PROMPTS for Restructuring Oral Muscular Phonetic Targets) will be evaluated from a behavioral and neuroanatomical point of view.

Objective: the current study is aimed to assess speech-language and white matter microstructure and volumetric changes induced by the PROMPT treatment.

Participants: Twenty-two Children with CAS aged 4 -12 years are enrolled and assigned to a PROMPT treatment (PROMPT-t ) or a Language and Non-Speech Oral Motor-treatment group (LNSOM-t).

Methods: All children with CAS will undergo a comprehensive clinical, neurological and speech-language assessment. The following procedures will be applied: a) anamnestic interview b) oral non verbal and verbal movements eveluation c) phonetic inventory, accuracy and consistency of speech d) DDK (Diadochokinetic rate, receptive and expressive vocabulary and grammar tests; f) spontaneous language analysis. These multiple measurements were aggregated and converted into a speech and language composite score.

MRI data will be acquired using a 1.5 T MR scanner. Structural images obtained with a 3D isotropic T1 weighted sequence will be analysed to evaluate volumetric alterations, to investigate cortical thickness and automatically delineate various Regions of Interest (ROIs). HARDI images will be acquired using 32 gradient directions and will be processed using tools available in FSL and MRtrix. Tract-based spatial statistics (TBSS) will be used to statistically analyse images of FA and mean diffusivity. Fiber tracts will be calculated using constrained spherical deconvolution and probabilistic tractography. Connectomes will be calculated by combining ROIs obtained from the structural images with tractography. Network-based analysis will be used to statistically analyse connectomes.

Speech and language assessment and brain MRI VBM and DTI analysis will be performed at baseline and at the end of the treatment.

Statistical analysis: Paired t-test on pre and post treatment behavioural and MRI/DTI measures will be performed to assess the changes within each of the two groups. Moreover, comparisons between the two groups at T0 and T1 will be performed by means of non parametric tests.

Evaluation of potentially training-induced changes of brain structural connectivity may provide further support to the hypothesis that CAS is due to a disruption of networks subserving the speech production system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic CAS based on the presence of specific diagnostic features of apraxia of speech (see ASHA and Strand et al's criteria) and on a comprehensive clinical and neurological assessment.
* Non-verbal IQ within the normal range at standardized tests of intelligence.
* Normal structural brain MRI.
* Acquisition of parents' informed consent to the execution of behavoiural and neuroradiological assessment at baseline and to perform speech/language treatment.

Exclusion Criteria:

* Orofacial structural abnormalities.
* Known pathologies of neurological, neurometabolical and genetic etiologies.
* Audiological deficits.
* Epilepsy.
* Intellectual disability.
* Autism spectrum disorder.

Ages: 4 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: 24 children with idiopathic CAS aged between 4 and 12 years. All the chidren are able to collaborate during MRI acquisition and behavioural assessment and to actively participate in the treatment sessions.
  To facilitate children's collaboration during MRI execution, a 0 Tesla simulator, reproducing the MRI setting of evaluation will be applied. Moreover during MRI acquisition children will be invited to watch cartoons through special glasses
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Speech Composite Severity Score changes after 7 months of treatment | At baselin and at 7 months of individual speech and language training
  Speech Severity Score aggregates measures of DDK, inaccuracy, inconsistency, Phonetic inventory, Syllable Omissions. Score ranges form: 0 (normal) to 5 (severely impaired)

SECONDARY OUTCOMES:
Post treatment Diffusion Weighed Imaging (DWI) metrics | At baseline and at 7 months of speech and language training
  Fractional Anisotropy (FA)
Post treatment Diffusion Weighed Imaging (DWI) changes | At baseline and at 7 months of speech and language training
  MD (Mean Diffusivity)
Post treatment cortical volumes modifications | At baseline and at 7 months of speech and language training
  Cortical thickness
Post treatment cortical volumes changes | At baseline and at 7 months of speech and language training
  Volumes analysis

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chilosi, Principal Investigator — IRCCS Stella Maris Foundation
Locations (1):
- IRCCS Fondazione Stella Maris, Tirrenia, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The results of each individual participant's evaluations will be coded and entered in a computerized database. Descriptive statistical analyses may be shared with other researchers on request .

REFERENCES:
- [Background] Kadis DS, Goshulak D, Namasivayam A, Pukonen M, Kroll R, De Nil LF, Pang EW, Lerch JP. Cortical thickness in children receiving intensive therapy for idiopathic apraxia of speech. Brain Topogr. 2014 Mar;27(2):240-7. doi: 10.1007/s10548-013-0308-8. Epub 2013 Aug 24. PMID 23974724
- [Background] Fiori S, Guzzetta A, Mitra J, Pannek K, Pasquariello R, Cipriani P, Tosetti M, Cioni G, Rose SE, Chilosi A. Neuroanatomical correlates of childhood apraxia of speech: A connectomic approach. Neuroimage Clin. 2016 Nov 4;12:894-901. doi: 10.1016/j.nicl.2016.11.003. eCollection 2016. PMID 27882295
- [Background] Square PA, Namasivayam AK, Bose A, Goshulak D, Hayden D. Multi-sensory treatment for children with developmental motor speech disorders. Int J Lang Commun Disord. 2014 Sep-Oct;49(5):527-42. doi: 10.1111/1460-6984.12083. Epub 2014 Mar 12. No abstract available. PMID 24617702
- [Background] Morgan AT, Su M, Reilly S, Conti-Ramsden G, Connelly A, Liegeois FJ. A Brain Marker for Developmental Speech Disorders. J Pediatr. 2018 Jul;198:234-239.e1. doi: 10.1016/j.jpeds.2018.02.043. Epub 2018 Apr 25. PMID 29705112
- [Background] Dale PS, Hayden DA. Treating speech subsystems in childhood apraxia of speech with tactual input: the PROMPT approach. Am J Speech Lang Pathol. 2013 Nov;22(4):644-61. doi: 10.1044/1058-0360(2013/12-0055). Epub 2013 Jun 28. PMID 23813194
- [Background] Namasivayam AK, Huynh A, Granata F, Law V, van Lieshout P. PROMPT intervention for children with severe speech motor delay: a randomized control trial. Pediatr Res. 2021 Feb;89(3):613-621. doi: 10.1038/s41390-020-0924-4. Epub 2020 May 1. PMID 32357364